CLINICAL TRIAL: NCT02121743
Title: Prospective, Multicenter, Randomized, Parallel Group Clinical Study Evaluating the Efficacy of a Biological Mesh (StratticeTM) for the Prevention of Parastomal Hernia After Colorectal Surgery With Colostomy
Brief Title: Use of a Biological Mesh (StratticeTM) for the Prevention of Parastomal Hernia After Colorectal Surgery With Colostomy
Acronym: PROBIOCOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI2014_843_0001; 2013-A01461-44 (Other: ID-RCB)
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Parastomal Hernia; Terminal Colostomy
Keywords: strattice; colostomy; parastomal hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strattice (Experimental): a strattice (10 x 10) will be used during the surgery, prior to the colostomy's conception
  Interventions: Device: strattice
- No strattice (Placebo Comparator): the colostomy is not reinforced with a mesh
  Interventions: Procedure: No strattice

INTERVENTIONS:
Device: strattice — use of a strattice
  Arms: Strattice
Procedure: No strattice — no use of a strattice
  Arms: No strattice

SUMMARY:
In France around 5,000 colostomies are performed after elective or emergency surgery. These colostomies could be associated with major outcomes including parastomal hernia (4 - 53%) of cases.

To reduce the incidence of these outcomes, several methods have been proposed but the more pertinent consist in the use of a biological mesh during the stoma's conception.

Nevertheless there is no data on the use of a biological mesh (StratticeTM) for the prevention of parastomal hernia.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a colorectal surgery with a terminal colostomy
* Elective or emergency surgery

Exclusion Criteria:

* Has collagen-vascular, connective tissue, or uncorrectable bleeding disorders as determined clinically by the PI.
* Has any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability.
* Has an autoimmune disease, an immune deficiency, or is on immune suppression drugs
* Is pregnant, or lactating.
* Allergic to any porcine or collagen products.
* survival < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
rate of parastomal hernia | postoperative month 6
  the presence of a parastomal hernia will be diagnosed either by the clinical examination either by a CT scan

SECONDARY OUTCOMES:
evaluation of the pain | 2 years after the surgery
  The pain will be evaluated with a visual scale 1 month, 6 months, 1 year and 2 years after the surgery
the postoperative morbidity | postoperative month 1
  the postoperative morbidity will be assessed with the Dindo Clavien classification
the parastomal hernia rate | postoperative year 1
  The parastomal hernia rate will be evaluated 1 year after the surgery during the clinical examination
the quality of life | 2 years after the surgery
  The quality of life will be assessed with the STOMA QoL form, the 12-Item Short Form Health Survey (SF12) and the Carolina comfort scale at 1 month, 6 months, 1 year and 2 years after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: jean marc regimbeau, MD, PhD, Principal Investigator — CHU Amiens
Locations (7):
- France (7):
  - Amiens Universitary Hospital, Amiens
  - Amiens university hospital, Amiens
  - Beauvais hospital, Beauvais
  - Caen hospital, Caen
  - Claude Huriet Hospital, Lille
  - Lariboisiere Hospital, Paris
  - Charles Nicolle Hospital, Rouen

REFERENCES:
- [Background] Timmermans L, Deerenberg EB, Lamme B, Jeekel J, Lange JF. Parastomal hernia is an independent risk factor for incisional hernia in patients with end colostomy. Surgery. 2014 Jan;155(1):178-83. doi: 10.1016/j.surg.2013.06.014. Epub 2013 Nov 12. PMID 24238119
- [Background] Lee L, Saleem A, Landry T, Latimer E, Chaudhury P, Feldman LS. Cost effectiveness of mesh prophylaxis to prevent parastomal hernia in patients undergoing permanent colostomy for rectal cancer. J Am Coll Surg. 2014 Jan;218(1):82-91. doi: 10.1016/j.jamcollsurg.2013.09.015. Epub 2013 Sep 29. PMID 24210147
- [Background] Swann JM, Turek FW. Transfer from long to short days reduces the frequency of pulsatile luteinizing hormone release in intact but not in castrated male golden hamsters. Neuroendocrinology. 1988 Apr;47(4):343-9. doi: 10.1159/000124935. PMID 3374759